CLINICAL TRIAL: NCT03705871
Title: Maxillary Expander With Differential Opening Versus Fan-type Expander: a Randomized Clinical Trial
Brief Title: Dentoskeletal Effects of the Expander With Differential Opening and the Fan-type Expander
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Camila Massaro, DDS, MSc and PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71648917.6.0000.5417
Record Dates: First submitted 2018-10-07; First posted 2018-10-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Malocclusion; Crossbite (Posterior)
Keywords: Palatal Expansion Technique; Cone-Beam Computed Tomography; Dental Models
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Differential Expansion Group (Experimental): The experimental group will be comprised 24 patients treated with a rapid maxillary expansion using the expander with differential opening. The expander is composed by two screws, one posteriorly and the other anteriorly positioned on the palate.
  Interventions: Device: Differential Expansion
- Fan-Fype Expander Group (Active Comparator): The active comparator group will be comprised by 24 patients treated with rapid maxillary expansion using the the fan-type expander. The expander is composed by one screw anteriorly positioned on the palate.
  Interventions: Device: Fan-Fype Expander

INTERVENTIONS:
Device: Differential Expansion — Twenty-four patients will be treated with a rapid maxillary expansion using the expander with differential opening. Appliance anchorage will be performed by bands adapted in the second maxillary deciduous molars and circumferential clamps will be bonded to the maxillary deciduous canines. The activation protocols will totalize an opening of 8mm in the anterior screw of the expander. After the active period of RME, the screws will be fixed with acrylic resin and the appliance will be kept as a retainer for 6 months.
  Arms: Differential Expansion Group
Device: Fan-Fype Expander — Twenty-four patients will be treated with a rapid maxillary expansion using the fan-type expander. Appliance anchorage will be performed by bands adapted in the second maxillary deciduous molars and circumferential clamps will be bonded to the maxillary deciduous canines. The activation protocols will totalize an opening of 8mm screw of the expander. After the active period of RME, the screws will be fixed with acrylic resin and the appliance will be kept as a retainer for 6 months.
  Arms: Fan-Fype Expander Group

SUMMARY:
This study will assess the dentoskeletal effects of two types of maxillary expanders in orthodontic patients in the mixed dentition, from 7 to 11 years old. Half of participants will be treated using the expander with differential opening, while the other half will undergo rapid maxillary expansion using the fan-type expander. The null hypothesis is that there is no difference between dentoskeletal effects of the two protocols.

DETAILED DESCRIPTION:
Rapid maxillary expansion (RME) is the orthopedic procedure of choice to treat maxillary constriction and posterior crossbite, and the study of dental, skeletal and periodontal effects of this procedure has been widely discussed in the orthodontic literature. The conventional RME expanders promote a similar expansion in the anterior and posterior regions of the maxillary arch. On the other hand, the fan-type expander allows the expansion concentrated in the intercanine region with little effects the intermolar distance. Finally, the expander with differential opening has two palatal screws and the differential activation protocol promotes a different amount of expansion for the anterior and posterior regions of the maxilla. No clinical study compared dental and skeletal effects of the expander with differential opening with those of the fan-type expander, including a three-dimensional analysis using CBCT exams and digital dental models. So, the aim of the present randomized clinical trial is to compare the skeletal and dentoalveolar effects of the maxillary expander with differential opening and the fan-type expander in the mixed dentition.

For this, patients will be recruited at the Orthodontic Clinic of Bauru Dental School, University of São Paulo, Brazil. A sample of 48 patients from 7 to 11 years old with transverse maxillary dental arch constriction will be prospectively and randomly allocated into two study groups. The first group will consist of 24 individuals treated with the expander with differential opening (DEG). The second group will consist of 24 individuals treated with the fan-type expander (FEG). In 12 patients from each group (immediate subgroups), a cone-beam computed tomography (CBCT) will be performed in the beginning of treatment (T1) and immediately after the rapid maxillary expansion (T2). In the other 24 patients, 12 from DEG and 12 from FEG (late subgroups), a CBCT will be obtained at T1 and 6 months after maxillary expansion (T3). Dental models will be obtained for all patients at T1 and T3. In digital dental models, maxillary arch width, perimeter, length and shape will be assessed. Standardized CBCT coronal sections will be used for measuring maxillary transverse dimensions, nasal cavity width and posterior tooth inclinations. Segmentation and superimposition of T1 and T3 CBCT images at the cranial base will be also performed. The opening of the midpalatal suture at the anterior and posterior region and the geometry of the suture opening will be evaluated in axial reconstructions of the CBCT.Discomfort, pain and quality of life will be evaluated by questionnaires.

After the normality test, the paired t test will be used in the intragroup comparison, and the independent t test will be used in the intergroup comparison. In the case of lost to follow-up patients, intention to treat analysis will be used. A significance level of 5% will be regarded for all tests.

Possible harms that could appear are related to temporary discomfort during the first days after the installation of the expander. Patients and legal guardians will be carefully oriented and they will be able to stop the treatment at any moment.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Mixed dentition;
* Ages ranging from 7 to 11 years old;
* Maxillary constriction associated to posterior crossbites;
* Angle Class I or Angle Class II malocclusions.

Exclusion Criteria:

* Cleft lip and palate;
* Craniofacial syndromes;
* Carious lesions;
* Angle Class III malocclusion;
* History of previous orthodontic treatment.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Maxillary and mandibular arch width (mm) | 6 months
  Measurements will be performed in digital dental models
Maxillary and mandibular arch length | 6 months
  Measurements will be performed in digital dental models
Maxillary and mandibular arch perimeter (mm) | 6 months
  Measurements will be performed in digital dental models
Nasal cavity width (mm) | 6 months
  Measurements will be performed in coronal sections of CBCT exams.
Maxillary width (mm) | 6 months
  Measurements will be performed in coronal sections of CBCT exams.
Maxillary molars inclination (°) | 6 months
  Measurement will be performed in CBCT scans.
Maxillary deciduous canines inclination (°) | 6 months
  Measurement be performed CBCT scans.
Amount of interincisor diastema (mm) | 10 days
  Measurement will be assessed in CBCT scans.
Opening of the midpalatal suture (mm) | 10 days
  Measurement be assessed in axial and coronal sections of CBCT scans.

SECONDARY OUTCOMES:
Discomfort evaluation using questionnaires | 1 month
  A Visual Analog Scale will be used from 0 to 10 cm.
Quality of life evaluation using questionnaires | 6 months
  The Child Perceptions Questionnaire (CPQ8-10) will be used to evaluate the quality of life of the patients before and after treatment.
Dentoskeletal displacements by three-dimensional superimposition of CBCT scams. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru Dental School - University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira R, Massaro C, Garib D. Vertical and sagittal changes produced by an expander with differential opening versus a fan-type expander: A post-hoc analysis of a randomised controlled trial. J Orthod. 2024 Dec;51(4):388-396. doi: 10.1177/14653125231208465. Epub 2023 Oct 31. PMID 37905906
- [Derived] Massaro C, Garib D, Cevidanes L, Janson G, Yatabe M, Lauris JRP, Ruellas AC. Maxillary dentoskeletal outcomes of the expander with differential opening and the fan-type expander: a randomized controlled trial. Clin Oral Investig. 2021 Sep;25(9):5247-5256. doi: 10.1007/s00784-021-03832-9. Epub 2021 Feb 12. PMID 33580351
- [Derived] Massaro C, Janson G, Miranda F, Aliaga-Del Castillo A, Pugliese F, Lauris JRP, Garib D. Dental arch changes comparison between expander with differential opening and fan-type expander: a randomized controlled trial. Eur J Orthod. 2021 Jun 8;43(3):265-273. doi: 10.1093/ejo/cjaa050. PMID 32840319